CLINICAL TRIAL: NCT04997135
Title: Clinical Evaluation of Therapeutic Meibomian Gland Expression
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-6455
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Visual Acuity; Meibomian Gland

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Meibography Subjects: Eligible subjects will undergo testing to evaluate the Meibomian gland appearance

SUMMARY:
This will be a single centre pilot study to evaluate appearance of the Meibomian glands.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be between 18 and 60 (inclusive) years of age at the time of screening. Inclusion Criteria at Baseline Evaluation.
  4. The subject must have visual acuity of 0.2 high contrast logMAR or better in their current correction or unaided in each eye.
  5. The subject must have at least 10 Meibomian glands yielding liquid secretion (MGYLS) in central lower eyelid region in each eye.
  6. The subject eyelids must be easy to evert, at the Investigator's discretion.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Be currently pregnant or breastfeeding.
  2. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g., rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See Section 9.1 for additional details regarding excluded systemic medications.
  3. Have any known hypersensitivity or allergic reaction to any of the known ingredients in the anesthetic (proxymetacaine hydrochloride) or sodium fluorescein.
  4. Have a history of cardiac disease or hyperthyroidism.
  5. Have had any previous ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, cataract etc.)
  6. Have participated in any ophthalmic clinical trial within 14 days prior to study enrolment.
  7. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  8. Have a history of amblyopia or strabismus.
  9. Have a history of contact lens wear. A trial period (up to one week) in the past is allowed.
  10. Wear eye makeup on the days of the study visits.
  11. Have clinically significant (grade 3 or higher on the Efron grading scale) slit lamp findings (e.g., corneal edema or neovascularization, conjunctival or limbal redness) or any other abnormality which would normally contraindicate participation in the study.
  12. Have any ocular infection.
  13. Have central lower eyelid Meibomian gland atrophy that exceeds 25%.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited and enrolled based on Inclusion/Exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Meibomian Gland Appearance | up to 2-week follow-up
  Meibomian gland appearance will be evaluated on both eyes using a custom image analysis algorithm, which calculates length ratio, width, area, intensity, tortuosity, and contrast

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu